CLINICAL TRIAL: NCT03303612
Title: Comparison of a Clinical Monitoring Strategy Versus Electrophysiology-guided Algorithmic Approach in Patients With a New Left Bundle Branch Block After Transcatheter Aortic Valve Implantation (TAVI) a Bayesian Randomized Trial (COME-TAVI)
Brief Title: Clinical Monitoring Strategy Versus Electrophysiology-guided Algorithmic Approach With a New LBBB After TAVI
Acronym: COME-TAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICM#2015-1949
Record Dates: First submitted 2016-05-06; First posted 2017-10-06 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Left Bundle-Branch Block; Aortic Valve Stenosis
MeSH Terms: conditions — Bundle-Branch Block; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EP-based approach/pacemaker implant (Other): Subjects will undergo an EP study prior to hospital discharge and will receive a pacemaker implantation if the HV interval is ≥65 msec.
  In the case where the electrical slowdown is not confirmed by the electrophysiological study, the participant will not have a pacemaker implantation.
  Interventions: Device: Pacemaker implant
- Compared transcutaneous cardiac monitor (Other): Subjects will undergo a minimum of 72 hour ECG monitoring in hospital and receive transcutaneous monitoring prior to hospital discharge for a duration of 30 days.
  Interventions: Device: Transcutaneous cardiac monitor

INTERVENTIONS:
Device: Pacemaker implant — Patient will be in the electrophysiology laboratory. The doctor will freeze the groin area and a medication may be given to help the patient relax. A catheter will be inserted into the groin up to the heart and the heart's electrical system will be recorded.
  Arms: EP-based approach/pacemaker implant
Device: Transcutaneous cardiac monitor — Transcutaneous cardiac patches will allow continuous electrocardiographic monitoring for a 30-day period. For the first randomized patients at the Montreal Heart Institute, Icentia was used and then was changed to a m-Health® device which allows continuous cardiac monitoring. The PocketECG from m-Health® is attached to 3 electrodes on the chest and contains a SIM card that transmits to a server located in Burlington, Ontario .The COME-TAVI coordinating center and the associated site will be informed rapidly of any events that occur . These events include:
  Ventricular fibrillation; Sustained ventricular tachycardia Any RR interval >5 sec; Third-degree AV block or Mobitz 2 AV block;
  Arms: Compared transcutaneous cardiac monitor

SUMMARY:
The primary hypothesis of the proposed study is that an electrophysiology-based algorithmic approach is superior to standard clinical follow-up with 30-day monitoring in reducing the combined endpoint of syncope, hospitalization, and death in patients in patients with new of left bundle branch block following transcatheter aortic valve implantation (TAVI).

DETAILED DESCRIPTION:
The study population consists of pacemaker-free patients that are 18 years or older undergoing a TAVI with new onset left bundle branch block. Patient consent is required.

Patients meeting the inclusion criteria will be randomized in a 1:1 ratio to one of the following two groups:

Group 1: electrophysiology-based algorithmic approach

Group 2: standard clinical follow-up with transcutaneous cardiac monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Informed consent to participate
* Persistent new-onset LBBB after TAVI implantation (i.e. present at day 2)

Exclusion Criteria:

* Prior pacemaker or implantable cardioverter-defibrillator
* Pre-existing right bundle branch block (RBBB) or LBBB (i.e., prior to TAVI)
* Class I or IIA indication for PPM implantation according to management guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-10-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with cardiovascular hospitalization, and/or syncope, and/or death after TAVI. | 12 months
  This is the number of participants who experienced cardiovascular hospitalizations, and/or syncope, and/or death after TAVI.

SECONDARY OUTCOMES:
Number of participants with cardiovascular hospitalizations. | 12 months
  This is the number of participants who were hospitalized for cardiovascular reasons within one-year post-TAVI.
Number of participants with hospitalisations (Total) | 12 months
  This is the number of participants who were hospitalized one-year post-TAVI.
Number of participants with emergency visits. | 12 months
  This is the number of participants who had emergency visits after TAVI.
Number of participants experiencing syncope | 12 months
  This is the number of participants who experienced syncope after TAVI.
Cost-effectiveness of EP-guided procedure compared to cardiac monitoring [incremental cost effectiveness ratio (ICER)]. | 12 months
  This is the incremental cost effectiveness ratio (ICER) for one strategy compared to the other.
Number of procedural complications in the group of EP-guided procedure compared to the group of cardiac monitoring. | 30 days
  This is the number of procedural complications in the group of EP-guided approach compared to cardiac monitoring within 30 days.
Number of atrio-ventricular blocks in the group of EP-guided procedure compared to the group of transcutaneous cardiac monitoring. | 12 months
  This is the number of atrio-ventricular blocks in the EP-guided procedure group compared to the transcutaneous cardiac monitoring group within 12 months of TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Léna Rivard, MD, MSC, Principal Investigator — Montreal Heart Institute
Locations (10):
- Canada (9):
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - New Brunswick Heart Center, Saint John, New Brunswick
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - London Health Sciences Center (LHSC), London, Ontario
  - University of Ottawa Heart Institute (UOHI), Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - CIUSSS du Nord de l'Île de Mtl, Montreal, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada
- Centre Hospitalier Universitaire de Nantes, Nantes, Cedex 01, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rivard L, Nault I, Krahn AD, Daneault B, Roux JF, Natarajan M, Healey JS, Quadros K, Sandhu RK, Kouz R, Greiss I, Leong-Sit P, Gourraud JB, Ben Ali W, Asgar A, Aguilar M, Bonan R, Cadrin-Tourigny J, Cartier R, Dorval JF, Dubuc M, Durrleman N, Dyrda K, Guerra P, Ibrahim M, Ibrahim R, Macle L, Mondesert B, Moss E, Raymond-Paquin A, Roy D, Tadros R, Thibault B, Talajic M, Nozza A, Guertin MC, Khairy P. Rationale and Design of the Randomized Bayesian Multicenter COME-TAVI Trial in Patients With a New Onset Left Bundle Branch Block. CJC Open. 2023 Jul 13;5(8):611-618. doi: 10.1016/j.cjco.2023.05.009. eCollection 2023 Aug. PMID 37720184